CLINICAL TRIAL: NCT05346159
Title: Effects of Adrenal Androgens on Gender-typed Behavior in Girls With Turner Syndrome
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Menatalla Moamen Ramadan Mohamed, resident doctor at pediatric department, Sohag University
Other Study IDs: soh-med-22-04-09
Record Dates: First submitted 2022-04-17; First posted 2022-04-26 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Turner Syndrome
MeSH Terms: conditions — Turner Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- turner syndrome group
  Interventions: Diagnostic Test: the correlation between level of adrenal androgen and gender-typed behavior in Girls with TS
- control group
  Interventions: Diagnostic Test: the correlation between level of adrenal androgen and gender-typed behavior in Girls with TS

INTERVENTIONS:
Diagnostic Test: the correlation between level of adrenal androgen and gender-typed behavior in Girls with TS — Laboratory assessment Serum dehydroepiandrosterone sulfate (DHEAS), follicle stimulating hormone (FSH), luteinizing hormone (LH) and estradiol (E2) will be measured using an enzyme mediated chemiluminescence for all participants Gender-typed behavior assessment
  * Parents of girls aged two to six years will evaluate their children's gender-typed behavior using the Pre school Activities Inventory
  * For girls above 6 years gender characteristics and gender role behavior will be evaluated using The Children's Sex Role Inventory (Child-adapted version of the original Bem Sex Role Inventory)
  * For all participants a Parent-Report Gender Identity Questionnaire for Children will be used to evaluate gender role behavior

SUMMARY:
Turner syndrome (TS) is a genetic disorder in which there is loss of all or part of the second X chromosome and occurs in 1/2500 live female births. TS is characterized by short stature and endocrine abnormalities, such as the loss of ovarian function (Gonadal dysgenesis) and estrogen deficiency.

The absence of pubertal development is one of the most common clinical features of patients with TS, who should have experienced a sex hormone surge if the hypothalamic-pituitary-gonadal axis was activated normally . Gonadarche and adrenarche are regarded as processes that are independent of each other. The function of adrenal gland is independent of true (central/complete/gonadotropin- dependent) puberty . Adrenal androgen in Turner syndrome shows a wide spectrum, ranging from normal to highly elevated.

X-linked genes affect the brain in at least two ways: by directly acting on the brain and by indirectly acting on the gonads to induce differences in specific gonadal secretions (i.e., hormones) that have specific effects on brain development. The changes in brain and behavioral/ cognitive phenotypes in TS individuals may be the result of a direct genetic factor, an indirect hormonal factor, or a combination of the two factors .

To evaluate direct effect of X chromosome, a lot of neuroimaging studies have revealed both neuroanatomical and neurofunctional changes in patients with TS. S. C. Mueller (2013) reported that oestrogen deficiency exhibits paradoxical healthy male-like patterns (i.e., a larger amygdala but reduced hippocampal volume). This finding confirms the indirect hormonal effect on the brain that are likely attributed to the effect of androgen on the brain or may be due to active role of estrogen in feminization of brain .

The cognitive phenotypes of TS include severe deficits in multiple cognitive domains: visual-spatial ability, mathematical processing, and social cognition. Regarding intelligence, numerous TS studies have a lower performance IQ in contrast to a within-normal verbal IQ in TS individuals .

The presence of hypogonadism with normal or may be elevated adrenal function in girls with turner syndrome provide a model to study the hormonal effect of adrenal androgen in absence of estrogen on gender-role behavior. Ehrhardt et al (1970) reported that Women with TS are described as clearly feminine in their behavior and interests .

To the best of our knowledge, there have been no previous studies on the correlation between level of adrenal androgen and gender-typed behavior in Girls with TS.

ELIGIBILITY:
Inclusion Criteria:

* Girls with turner syndrome (TS) (karyotype 45, X) younger than 18 years of age and Tanner stage matched healthy control girls with normal karyotype attending outpatient clinic at Sohag University Hospital will be included in the study.

Exclusion Criteria:

* failure to obtain informed consent

Max Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Study Population: Girls with turner syndrome (TS) (karyotype 45, X) younger than 18 years of age and Tanner stage matched healthy control girls with normal karyotype attending outpatient clinic at Sohag University Hospital will be included in the study
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Serum dehydroepiandrosterone sulfate (DHEAS) | Baseline
  we use DHEAS level to access adrenal function
follicle stimulating hormone (FSH) | Baseline
  to access ovarian function
luteinizing hormone (LH) | Baseline
  to access ovarian function
estradiol (E2) | Baseline
  to access ovarian function
Gender-typed behavior | Baseline
  we will measure children's gender-typed behavior using the Pre school Activities Inventory
Gender-typed behavior The Children's Sex Role Inventory | Baseline
  we will measure children's gender-typed behavior using The Children's Sex Role Inventory
Parent-Report Gender Identity Questionnaire | Baseline
  we will measure children's gender-typed behavior using the Parent-Report Gender Identity Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Li M, Zhao C, Xie S, Liu X, Zhao Q, Zhang Z, Gong G. Effects of hypogonadism on brain development during adolescence in girls with Turner syndrome. Hum Brain Mapp. 2019 Dec 1;40(17):4901-4911. doi: 10.1002/hbm.24745. Epub 2019 Aug 7. PMID 31389646
- [Background] Counts DR, Pescovitz OH, Barnes KM, Hench KD, Chrousos GP, Sherins RJ, Comite F, Loriaux DL, Cutler GB Jr. Dissociation of adrenarche and gonadarche in precocious puberty and in isolated hypogonadotropic hypogonadism. J Clin Endocrinol Metab. 1987 Jun;64(6):1174-8. doi: 10.1210/jcem-64-6-1174. PMID 3571422
- [Background] Zhao C, Gong G. Mapping the effect of the X chromosome on the human brain: Neuroimaging evidence from Turner syndrome. Neurosci Biobehav Rev. 2017 Sep;80:263-275. doi: 10.1016/j.neubiorev.2017.05.023. Epub 2017 Jun 4. PMID 28591595
- [Background] Ehrhardt AA, Greenberg N, Money J. Female gender identity and absence of fetal gonadal hormones: Turner's syndrome. Johns Hopkins Med J. 1970 May;126(5):237-48. No abstract available. PMID 4911705
- [Background] Mueller SC. Magnetic resonance imaging in paediatric psychoneuroendocrinology: a new frontier for understanding the impact of hormones on emotion and cognition. J Neuroendocrinol. 2013 Aug;25(8):762-70. doi: 10.1111/jne.12048. PMID 23656557
- [Background] Johnson LL, Bradley SJ, Birkenfeld-Adams AS, Kuksis MA, Maing DM, Mitchell JN, Zucker KJ. A parent-report gender identity questionnaire for children. Arch Sex Behav. 2004 Apr;33(2):105-16. doi: 10.1023/b:aseb.0000014325.68094.f3. PMID 15146143
- [Background] Dorr HG, Penger T, Marx M, Rauh M, Oppelt PG, Volkl TKM. Adrenarche and pubarche in girls with turner syndrome during growth-promoting therapy with human growth hormone. BMC Endocr Disord. 2019 Jan 18;19(1):9. doi: 10.1186/s12902-019-0333-z. PMID 30658614